CLINICAL TRIAL: NCT05193890
Title: The Performance of Next-generation Sequencing in the Diagnosis of Epilepsy and/or Intellectual Disability in the Pediatric Cohort of the Regional University Hospital Center of Nancy
Brief Title: Using Next-generation Sequencing in the Diagnosis of Epilepsy and/or Intellectual Disability in a Pediatric Cohorte
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, calina TODOSI, MD, Pediatric Neurology, Central Hospital, Nancy, France
Other Study IDs: 2021PI127.
Record Dates: First submitted 2021-09-14; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Epilepsy; Intellectual Disability
MeSH Terms: conditions — Epilepsy; Intellectual Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epilepsy only: Epilepsy only patients who underwent our gene panel and the Clinical exome Solution
  Interventions: Genetic: retrospective analysis of a panel result
- Intelectual Disability only: Intelectual Disability only patients who underwent our gene panel and the Clinical exome Solution
  Interventions: Genetic: retrospective analysis of a panel result
- Epilepsy and Intelectual Disability: Intelectual Disability and Epilepsy patients who underwent our gene panel and the Clinical exome Solution
  Interventions: Genetic: retrospective analysis of a panel result

INTERVENTIONS:
Genetic: retrospective analysis of a panel result — retrospective analysis of a exome clinical solution

SUMMARY:
ABSTRACT

Background and Aims:

To determine the diagnostic performance of the epilepsy and intellectual disability panel used in the pediatric population, starting in June 2019, at the Regional University Hospital Center of Nancy, France.

Design:

An observational and retrospective study, at the Regional University Hospital Center of Nancy, France.

Materials and Methods:

Pediatric patients who underwent genetic analysis with the epilepsy-intellectual disability gene panel. All of these patients were either epileptic or had intellectual disability, or both, of undetermined etiology.

Results:

We included 69 patients in this study. We identified causative mutations in 46.4% (32 of 69 patients) of this cohort after the gene panel and 52.2% (36 patients) including positive results after realization of the Clinical Exome Solution.

DETAILED DESCRIPTION:
Epilepsy and intellectual disability are common and highly heterogeneous neurodevelopmental disorders in children. Their respective prevalence are 3.2 to 5.1/1000 (1,2) and 1.3 to 2.2% (3).

An epileptic seizure is due to abnormal excessive or synchronous neuronal activity. Epilepsy is defined by : (A) At least two unprovoked (or reflex) seizures occurring >24 h apart; or (B) one unprovoked (or reflex) seizure and a probability of further seizures at least 60% ; or (C) diagnosis of an epilepsy syndrome (4). Intellectual disability (ID) is defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), as a significant limitation in intellectual functioning and adaptive behavior, which include conceptual, social, and practical skills, arising before age 18.

These two conditions can be caused by a variety of environmental and genetic factors, often combined, making the diagnosis difficult (5,6). Standard diagnostic approaches include biochemical and enzyme analysis for neurometabolic disorders, MRI brain imaging and genome-wide microarray analysis (7-9).

Because of the large variability of genotypic-phenotypic expression (a syndrome can have several genetic causes; the same gene can be expressed in different ways) and the huge genetic heterogeneity, the identification of the genes involved in these pathologies has long been difficult. In recent decades, considerable progress has been made in genetics, with the development of new technologies such as next-generation sequencing (NGS). These new techniques permit the sequencing of many genes at the same time, at an ever lower cost, allowing the use of these tests in clinical practice routine with gene panels, and even whole-exome or whole-genome sequencing (10). We now identified more than 1000 genes implicated in mechanisms of epilepsy and ID, with various pathways (11-16).

ELIGIBILITY:
Inclusion Criteria:

* We included in our study all pediatric patients who underwent genetic analysis with the epilepsy-intellectual disability gene panel between June 2019 and May 2021. All of these patients were either epileptic or had intellectual disability, or both, of undetermined or genetic presumed etiology.

Exclusion Criteria:

* We excluded i) patients older than 18 years, ii) those for whom the indication for genetic analysis was not epilepsy or intellectual disability iii) patients not followed up at the Regional University Hospital Center of Nancy, France.

Ages: 1 Day to 17 Years | Sex: All
Age Groups: Child
Study Population: Of the 69 patients included in the study, the majority were boys, 62.3% (43 patients) and 37.7% were girls (26 patients). This difference is most pronounced in the subcategory of patients with intellectual disabilities, with a sex ratio of approximately 1:2,3. The median age of the population at inclusion was 5 years [2.2-17].
  From the total of 69 patients included in our study, the majority beneficiated of the gene panel for their intellectual disability (37 patients i.e. 53.6%), 13 for their epilepsy (18.8% of the patients) and 19 patients had both (i.e. 27.5%).
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
determine the pourcentage of positive résults using our epilepsy and intellectual disability panel | 2 years
  the pourcentage of positive résultats after the panel analysis

SECONDARY OUTCOMES:
evaluation of supplementary positive results of the CES | 2 years
  the pourcentage of positive résultats found using the CES and witch were negatif using the panel

CONTACTS AND LOCATIONS:
Locations (1):
- Calina Todosi, Vandœuvre-lès-Nancy, France